CLINICAL TRIAL: NCT03449043
Title: ANALYSIS OF THE BECOME OF THE PATIENTS ADDRESSED BY THEIR GENERAL PRACTITIONER TO EMERGENCIES OF UHC POITIERS
Brief Title: BECOME PATIENTS IN THE EMERGENCIES OF UHC POITIERS
Acronym: DEPAUG
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DEPAUG
Record Dates: First submitted 2018-02-19; First posted 2018-02-28 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-02

CONDITIONS: Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Real care course — Evaluate the rate of adequacy between the request made by the general practitioner and the response to emergencies

SUMMARY:
The number of consultations in the emergency services has continued to increase with 19.7 million passages in 2014, an increase of 4% compared to 2013. Among these admissions, many patients come spontaneously to the emergency department and others are sent by the general practitioner who remains the first resort in the care of the patient.

Faced with this massive influx to emergency services, the investigator will see what is the future of these. Are they more likely to be hospitalized than patients presenting to emergencies on their own?

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* View by a general practitioner whether he is their doctor or a substitute
* Addressed with a mail
* All types of pathologies are taken into account

Exclusion Criteria:

* Minor patient

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient coming to emergency for all types of pathologies with general practitioner letter
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Concordance rate between the general practitioner request and the patient's actual care path. | 1 day
  Medical file